CLINICAL TRIAL: NCT06809946
Title: Feasibility of Fluorescence Imaging with Bevaci-zumab-800CW During Bronchoscopy in Patients with a Pulmonary Lesion Considered to Be Malignant
Brief Title: Feasibility of Fluorescence Imaging with Bevacizumab-800CW During Bronchoscopy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 202100285; 2024-510793-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Lung Neoplasms; Pulmonary Neoplasms; Lymph Node Involvement
MeSH Terms: conditions — Lung Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluorescence molecular imaging arm with bevacizumab-800CW at dose of 15 mg (Active Comparator)
  Interventions: Drug: injection with 15 mg bevacizumab-800CW before bronchoscopy
- Fluorescence molecular imaging arm with bevacizumab-800CW at dose of 25 mg (Active Comparator)
  Interventions: Drug: injection with 25 mg bevacizumab-800CW before bronchoscopy

INTERVENTIONS:
Drug: injection with 15 mg bevacizumab-800CW before bronchoscopy — Patients will receive an intravenous administration of 15 mg bevacizumab-800CW before the bronchoscopy procedure. The bronchoscopy will start with high-definition white light bronchoscopy, followed by fluorescence molecular bronchoscoy to observe the fluorescence signal and MDSFR-SFF spectroscopy to quantify the fluores-cence signal in vivo.
  Arms: Fluorescence molecular imaging arm with bevacizumab-800CW at dose of 15 mg
Drug: injection with 25 mg bevacizumab-800CW before bronchoscopy — Patients will receive an intravenous administration of 15 mg bevacizumab-800CW before the bronchoscopy procedure. The bronchoscopy will start with high-definition white light bronchoscopy, followed by fluorescence molecular bronchoscoy to observe the fluorescence signal and MDSFR-SFF spectroscopy to quantify the fluores-cence signal in vivo.
  Arms: Fluorescence molecular imaging arm with bevacizumab-800CW at dose of 25 mg

SUMMARY:
In this feasibility study, bronchoscopy will be combined with fluorescence molecular imaging using the near-infrared fluorescence (NIRF) tracer bevacizumab-800CW for assessment of pulmonary lesions and/or lymph nodes considered to be malignant.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to participation in the study.
2. Age ≥ 18 years.
3. Patient has at least one intrabronchial, near-to-airway located or peripheral pulmonary nodule - with or without pathological lymph nodes - which is considered malignant (independent of its primary origin).
4. Patient is considered fit to undergo a diagnostic and/or therapeutic bronchoscopy (with or without addition of virtual navigation and/or endobronchial ultrasound; including propofol sedation or general anesthesia if either is indicated) to obtain tumor material according to standard care protocols.

Exclusion Criteria:

1. History of infusion reactions to bevacizumab.
2. Medical or psychiatric conditions that compromise the patient's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
In vivo fluorescent signal of malignant lesion versus non-tumorous tissue | Assessed directly during the bronchoscopy procedure